CLINICAL TRIAL: NCT07077837
Title: Effect of Incorporating Perceptual Learning Into Plantar Hardness Discrimination on the Risk of Falling and Muscle Torque in Patients With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hemiplegia
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hemiparesis; Balance
Keywords: planter pressure; hemiplegia; balance
MeSH Terms: conditions — Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received perceptual learning using plantar hardness discrimination and conventional treatmen
  Interventions: Other: Study Group
- control group (Active Comparator): received conventional treatment (balance exercise functional care training)
  Interventions: Other: Control

INTERVENTIONS:
Other: Study Group — received perceptual learning using plantar hardness discrimination and conventional treatment
  Arms: study group
Other: Control — received conventional treatment (balance exercise functional care training
  Arms: control group

SUMMARY:
Hemiplegia, a common stroke sequela, significantly impairs motor function, leading to balance issues and increased fall risk. Traditional rehabilitation methods often fall short in fully restoring function. This study explores Perceptual Learning's role in enhancing balance training outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • age from 45 to 65 years old

  * both Sex
  * the duration of illness more than six months
  * post stroke hemiplegia
  * spasticity ranged from (1:1+) according to Modified Ashworth Scale
  * Body mass index (BMI) ranged from 18.5 to 29.9 Kg/m2.

Exclusion Criteria:

* 1) stroke occurred less than 3 months ago (2) Patients with severe cognitive or psychiatric impairment aphasia who could not understand the instructions given to him by physical therapist or unable to perform the task (3) any other orthopedic disorders or neurologic diseases.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
risk of fall | 4 weeks
  The Biodex Balance System is advice to measure different parameter of body balance, posture stability and risk of falling

SECONDARY OUTCOMES:
muscle torque | 4 weeks
  Isokinetic devices are used in assessments to evaluate muscle strength and function by measuring resistance at a constant speed. These devices, often called isokinetic dynamometers, are particularly helpful in identifying muscle weaknesses
Functional independent measures scale | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No